CLINICAL TRIAL: NCT05953558
Title: Cohorte Française Des Patients Implantés de Micra AV
Brief Title: French Cohort Evaluating the effectiveneSs of Atrioventricular Synchrony by the micRa AV
Acronym: AV-CESAR
Status: Recruiting | Type: Observational
Sponsor: Paris Sudden Death Expertise Center (Other)
Collaborators: CHU de Tours (Unknown); European Georges Pompidou Hospital (Other); Hôpital privé Clairval - Marseille (Unknown); Clinique Pasteur Toulouse (Other); University Hospital, Bordeaux (Other); Infirmerie Protestante Lyon (Ambiguous); Institut Jacques Cartier - Massy (Unknown); University Hospital, Grenoble (Other); Hôpital de la Timone (Other); University Hospital, Toulouse (Other); Hopital Prive Saint Martin - Bordeaux (Unknown); Hospices Civils de Lyon (Other); CHU de Rouen - Accueil (Other); University Hospital, Caen (Other); Médipôle Lyon-Villeurbanne (Other); Hospital Ambroise Paré Paris (Other); Clinique Saint Augustin - Bordeaux (Unknown); Rennes University Hospital (Other); Clinique de la Sauvegarde - Lyon (Unknown); University Hospital of Saint-Etienne (Other); Hôpital Privé de Parly II - Le Chesnay (Other); Institut Mutualiste Montsouris (Other); Centre Hospitalier Universitaire, Amiens (Other); University Hospital, Clermont-Ferrand (Other); Centre Hospitalier Régional et Universitaire de Brest (Other); Poitiers University Hospital (Other); Clinique Saint-Gatien - Tours (Unknown); CHU de Reims (Other); Centre Hospitalier Universitaire de Besancon (Other); Centre Hospitalier Universitaire Dijon (Other); Hôpital Privé de Lille Métropole (Unknown); University Hospital, Montpellier (Other); University Hospital, Strasbourg, France (Other); Nantes University Hospital (Other); Centre Cardio-Thoracique de Monaco (Unknown); Hospital St. Joseph, Marseille, France (Other); Centre Hospitalier Régional Metz-Thionville (Other); Centre Hospitalier Annecy Genevois (Other); Clinique du Millenaire (Other); University Hospital, Limoges (Other); Clinique Saint Pierre - Perpignan (Unknown); Bichat Hospital (Other); Universite de La Reunion (Other); CHU de Lille (Unknown); Institute Arnault Tzanck, France (Other); Hôpital Privé Les Franciscaines (Other); CHU de Fort de France - Martinique (Unknown); Henri Mondor University Hospital (Other); University Hospital, Angers (Other Government); Centre Hospitalier de Lens (Other); Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A00023-42 Protocole
Record Dates: First submitted 2023-06-21; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Atrioventricular Synchrony by the Micra AV
Keywords: Pacemaker syndrome; Dual chamber pacemaker upgrade; Quality of life; SF36 questionnaire; Effectiveness; Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Patients implanted with Micra AV — The first 1000 patients implanted by the device in France

SUMMARY:
Transvenous cardiac pacemakers have pitfalls due to lead- and device pocket-related complications. Leadless pacemakers were developed and introduced into clinical practice to overcome the weaknesses of traditional transvenous pacemakers. The absence of atrial pacing has restricted their uses mainly for cases of paroxysmal atrioventricular block (AVB) or AVB with atrial fibrillation. The Micra AV contains an embedded accelerometer that senses the atrial contraction waveform, allowing the ventricle to be paced once the atrial contraction is complete. This atrioventricular synchronization is intended to extend the use of the device to cases of permanent complete AVB with normal sinus function. Two randomized clinicals trials have been proven it's efficacy. However, with AV-CESAR cohort, we aim to evaluate the real word effectiveness of Micra AV, in the first 1000 patients implanted by the device in France.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent Micra AV implantation

Exclusion Criteria:

* Refusal of consent

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The first 1000 patients implanted with Micra AV in France since May 29, 2020
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Profile of patients implanted with Micra AV | Through study completion, an average of 3 years
  Description of the population of patients implanted by the device : age, sex, comorbidities (rate of hypertension, diabetes, ischemic heart disease, heart failure, severe pulmonary disease, severe chronic renal failure, cirrhosis, severe impairement of mobility, severe psychiatric disease or demencia and TAVR)
Follow-up occurrence of upgrading to a dual-chamber pacemaker | Through study completion, an average of 3 years
  Rate of pacemaker syndrome and requirement of dual-chamber pacemaker upgrade
Early and late device-related complications | Through study completion, an average of 3 years
  Rate of inhospital and late complications related to Micra AV

SECONDARY OUTCOMES:
Assessment of the quality of life in permanent atrioventricular block and normal sinus function subgroup | Through study completion, an average of 3 years
  Evaluation of the quality of life using the 36-item Short Form (SF-36) questionnaire in the subgroup of 150 patients implanted for permanent atrioventricular block and normal sinus function. SF-36 is a self-report questionnaire and composed of eight multi-item scales (Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, Mental Health), with scores for each of these scales ranging from 0 to 100. Higher scores indicate better health status. A mean score of 50 has been articulated as a normative value for all scales. The SF-36 has been translated and validated in French language.
Risk factors of a compromised quality of life | Through study completion, an average of 3 years
  Identify the risk factors associated with impaired quality of life in patients with Micra AV

CONTACTS AND LOCATIONS:
Overall Officials: Eloi Marijon, MD,PhD, Principal Investigator — Paris Sudden Death Expertise Center; Fawzi Kerkouri, MD, Principal Investigator — University hospital of Brest
Locations (1):
- Paris Cardiovascular Research Centre (AV-CESAR Investigators), Paris, France

IPD SHARING:
Plan to Share IPD: Undecided